CLINICAL TRIAL: NCT01933659
Title: Anti-bacterial Effects of Ingesting Deep Sea Water in Subjects With H. Pylori Infection
Brief Title: Anti-H. Pylori Effect of Deep See Water
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201304065RIND
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; deep see water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A: DSW group (Experimental): ingesting DSW 200 cc four times a day (one hour before meal and bed time);
  Interventions: Drug: DSW
- group B: non-DSW group (Placebo Comparator): ingesting non-DSW drinking water 200 cc four times a day (one hour before meal and bed time).

INTERVENTIONS:
Drug: DSW — ingesting DSW 200 cc four times a day (one hour before meal and bed time)
  Arms: group A: DSW group

SUMMARY:
Deep sea water (DSW) is characterized by high purity, low temperature, high nutrients and minerals and is obtained from the water flows 200 meters under the surface of the sea. The inhibition of H. pylori growth by DSW has been demonstrated in vitro study. However, up to now, there is few randomized control study to evaluate the anti-bacterial effects of ingesting DSW in patients with H. pylori infection.

The aims of this study are:

1. to evaluate the anti-bacterial effects of ingesting DSW in patients with H. pylori infection;
2. to evaluate the patient adherence and adverse effects of ingesting DSW.

DETAILED DESCRIPTION:
Patients having H. pylori-positive chronic gastritis with/without small erosions or peptic ulcer scars will be recruited. Before treatment, H. pylori infection status will be examined by endoscopy with biopsy or 13C-urea breath test (13C-UBT). All patients will receive 13C-UBT before treatment, at the end of 2 week's treatment and 4 weeks after termination of treatment. A computed generated random numbers sequence will be blocked (2:1; block sizes of six) into two groups, say A and B.

group A - ingesting DSW 200 cc four times a day (one hour before meal and bed time); group B - ingesting non-DSW drinking water 200 cc four times a day (one hour before meal and bed time).

To keep the study in double-blind model, the picture of package for DSW and non-DSW drinking water will be the same.

Prokinetics (metoclopramide 5 mg/tab 1 tid) and antacid (strocain tablet (oxethazaine 5 mg and polymigel 244 mg/tab) 1 tid) will be permitted for relieving the dyspeptic symptoms.

All patients will be asked to complete a questionnaire and to record symptoms and water/drug consumption daily during the treatment period. Post-treatment, the patients will be seen at the Outpatients Clinic to investigate patient adherence and adverse of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients having H. pylori-positive chronic gastritis with/without small erosions or peptic ulcer scars who are aged greater than 20 years and are willing to received anti-H. pylori treatment.

Exclusion Criteria:

* pregnant or nursing woman
* serious concomitant illness and malignant tumor of any kind
* serious bleeding from gastrointestinal tract
* previous gastric surgery
* receiving bismuth salts, Proton pump inhibitors, or antibiotics in the previous month.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
to compare the efficacy of DSW and non-DSW drinking water as anti-H. pylori regimen | 6 months
  The eradication rates (efficacy) will be evaluated by intention-to-treat (ITT) and per-protocol (PP) analysis.

SECONDARY OUTCOMES:
to compare the adverse effects and patient adherence of DSW and non-DSW drinking water as anti-H. pylori regimen | 6 months
  The safety and patient adherence will be evaluated by the number of participant with adverse events and by counting unused medication after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D.Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan